CLINICAL TRIAL: NCT06178198
Title: An Open-label, Single-arm, Single-center Clinical Trial to Evaluate the Efficacy and Safety of Yttrium-90 Ablative Radioembolization (Radiation Major Hepatectomy) for Unifocal Large Hepatocellular Carcinoma
Brief Title: Radiation Major Hepatectomy to Selectively Treat Large Unifocal Hepatocellular Carcinoma
Acronym: RESCUE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Woo Choi, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-2306-208-1446; NRF-2023R1A2C1006509 (Other Grant/Funding Number: National Research Fund of Korea)
Record Dates: First submitted 2023-11-30; First posted 2023-12-20 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Radioembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Open-label, prospective, single-arm, single-center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ablative radioembolization for large HCC (Experimental): Yttrium-90 resin microspheres (SIR-Sphere, SIRTEX) will be administered to cover the main tumor, satellite nodules, and margin.
  Interventions: Procedure: Ablative radioembolization using Yttrium-90 resin microspheres

INTERVENTIONS:
Procedure: Ablative radioembolization using Yttrium-90 resin microspheres — Based on 99mTc-MAA mapping, a partition model (multi-compartment MIRD) is employed to plan for a radiation dose of 400 (± 30%) to the tumor. If delivering this dose to the tumor is challenging due to lung dose limitations, the maximum feasible dose is administered to the tumor while maintaining the estimated lung dose below 15 Gy. While treating the entire tumor with a single high-dose radioembolization session is preferred, if necessary due to considerations like estimated lung dose, the treatment can be divided into two sessions, keeping the cumulative lung dose below 25 Gy. For any methods not covered in this discussion, refer to the SIR-Sphere user manual by Sirtex.

SUMMARY:
The RESCUE trial is a prospective, single-arm clinical study to evaluate the efficacy and safety of ablative radioembolization using Yttrium-90. This treatment is being investigated as a potential curative approach, as well as a bridging or downstaging strategy for surgery, in patients with large hepatocellular carcinoma (greater than 8 cm) who maintain good liver function.

DETAILED DESCRIPTION:
Patients presenting with large hepatocellular carcinoma (greater than 8 cm), whether accompanied by satellite nodules or not, but retaining good liver function, will undergo ablative radioembolization utilizing Yttrium-90 resin microspheres. This approach is designed to deliver an ablative dose to both tumors and the surrounding liver (i.e., margin) with curative intent, while preserving over 30% of the non-tumorous liver volume. The efficacy and safety of this treatment will be evaluated over a period of two years and 90 days, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and over.
2. Patients diagnosed with hepatocellular carcinoma histologically and/or radiologically (LI-RADS 4 or 5).
3. Patients with no more than five lesions in dynamic contrast-enhanced CT or MRI, and the largest tumor diameter exceeding 8 cm.
4. Patients without vascular invasion and bile duct invasion in dynamic contrast-enhanced CT or MRI.
5. Patients with no extrahepatic metastasis in lung CT and contrast-enhanced abdominal CT or MRI.
6. Patients with no prior treatment for liver cancer.
7. Child-Pugh class A.
8. ECOG performance status of 1 or less.
9. Patients with no major organ dysfunction according to blood tests performed within one month of study enrollment.

   1. Leukocytes ≥ 2,500/µL and ≤ 12,000/µL
   2. Absolute neutrophil count ≥ 1,500 /mm^3
   3. Hemoglobin ≥ 8.0 g/dL (transfusion allowed to meet this criterion)
   4. Total bilirubin ≤ 3.0 mg/dL
   5. Platelet ≥ 50,000/µL
   6. INR ≤ 2.0 for patients not taking anticoagulants
   7. AST ≤ 200 IU/L (i.e., ≤ 5X upper normal limit)
   8. ALT ≤ 200 IU/L (i.e., ≤ 5X upper normal limit)
   9. ALP ≤ 575 IU/L (i.e., ≤ 5X upper normal limit)
   10. Creatinine ≤ 2.0 mg/dL
10. Patients with a life expectancy of more than 3 months.
11. Patients who have adequately understood the clinical trial and consented in writing.
12. Non-pregnant women of childbearing potential.

Exclusion Criteria:

1. Patients who are not suitable for ablative radioembolization as indicated by pre-treatment testing with macro-aggregated albumin labeled with technetium-99 (99mTc-MAA) for radioembolization.

   1. Cases where the estimated lung dose exceeds 15 Gy when 150 Gy of absorbed dose is administered to the tumor based on the partition method.
   2. Cases with severe hepatic artery-portal vein shunting that might lead to irradiation of the non-tumorous liver segments.
2. Patients whose volume of non-tumorous liver not included in the treatment area is less than 30% of the total non-tumorous liver volume.
3. Patients scheduled to use immunotherapy irrespective of the response to radioembolization.
4. Patients who have had active cancer within the last two years prior to the clinical trial participation.
5. Patients who have undergone surgery or procedures related to the bile duct.
6. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate according to localized mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  The number of patients with partial or complete response as the best local response divided by the total number of participants
Duration of response according to localized mRECIST | Time of response up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  The time from first documentation of partial or complete response to the first documentation of progressive disease, death due to any cause, or receipt of subsequent anticancer treatment, whichever comes first

SECONDARY OUTCOMES:
Objective response rate according to mRECIST. | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Duration of response according to mRECIST | Time of response up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
2-year restricted mean duration of response according to localized mRECIST and mRECIST | Time of response up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or 24 months after the initial treatment
Complete response rate according to localized mRECIST and mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Duration of complete response according to localized mRECIST and mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
2-year restricted mean DoCR (RMDoCR) according to localized mRECIST and mRECIST | Time of complete response up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or 24 months after the initial treatment
Best response within 2-years according to localized mRECIST and mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Time to best response according to localized mRECIST and mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Time to progression according to localized mRECIST and mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Overall survival | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
2-year restricted mean survival time of overall survival | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or 24 months the initial treatment
Progression-free survival | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Hepatic progression-free survival (HPFS) | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Pathological necrosis rate (%) after curative resection or liver transplantation | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Time to subsequent HCC treatment | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Reason for subsequent HCC treatment | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Rate for conversion to curative resection and liver transplantation | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Adverse event and serious adverse event | Time of treatment up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
  Common Terminology Criteria for Adverse Events v5.0
Changes in Child-Pugh class | Baseline up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
Changes in ALBI (albumin-bilirubin) grade | Baseline up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
Changes in MELD (model for end-stage liver disease) score | Baseline up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
Changes in ECOG (Eastern Cooperative Oncology Group) performance status scale | Baseline up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
  0 (fully active) to 5 (dead)
Changes in health-related quality of life | Baseline up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
  EORTC QLQ-C30 and HCC18
Changes in regional liver function | Baseline up to 180 days after the initial treatment or subsequent anticancer treatment, whichever comes first
  99mTc-MAA hepatobiliary scan with SPECT-CT

OTHER OUTCOMES:
Pre-treatment dosimetry based on 99mTc-MAA SPECT-CT | Baseline
Post-treatment dosimetry based on Y90 PET-CT | Within two days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jin Woo Choi, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garin E, Tselikas L, Guiu B, Chalaye J, Edeline J, de Baere T, Assenat E, Tacher V, Robert C, Terroir-Cassou-Mounat M, Mariano-Goulart D, Amaddeo G, Palard X, Hollebecque A, Kafrouni M, Regnault H, Boudjema K, Grimaldi S, Fourcade M, Kobeiter H, Vibert E, Le Sourd S, Piron L, Sommacale D, Laffont S, Campillo-Gimenez B, Rolland Y; DOSISPHERE-01 Study Group. Personalised versus standard dosimetry approach of selective internal radiation therapy in patients with locally advanced hepatocellular carcinoma (DOSISPHERE-01): a randomised, multicentre, open-label phase 2 trial. Lancet Gastroenterol Hepatol. 2021 Jan;6(1):17-29. doi: 10.1016/S2468-1253(20)30290-9. Epub 2020 Nov 7. PMID 33166497
- [Background] Choi JW, Suh M, Paeng JC, Kim JH, Kim HC. Radiation Major Hepatectomy Using Ablative Dose Yttrium-90 Radioembolization in Patients with Hepatocellular Carcinoma 5 cm or Larger. J Vasc Interv Radiol. 2024 Feb;35(2):203-212. doi: 10.1016/j.jvir.2023.10.011. Epub 2023 Oct 21. PMID 37866475
- [Background] Levillain H, Bagni O, Deroose CM, Dieudonne A, Gnesin S, Grosser OS, Kappadath SC, Kennedy A, Kokabi N, Liu DM, Madoff DC, Mahvash A, Martinez de la Cuesta A, Ng DCE, Paprottka PM, Pettinato C, Rodriguez-Fraile M, Salem R, Sangro B, Strigari L, Sze DY, de Wit van der Veen BJ, Flamen P. International recommendations for personalised selective internal radiation therapy of primary and metastatic liver diseases with yttrium-90 resin microspheres. Eur J Nucl Med Mol Imaging. 2021 May;48(5):1570-1584. doi: 10.1007/s00259-020-05163-5. Epub 2021 Jan 12. PMID 33433699